CLINICAL TRIAL: NCT06879574
Title: Investigating a Data-driven Standardized and Objective Dietary Intake Assessment Tool in Free-living Individuals - SODIAT-2 Study
Brief Title: Identifying the Best Tools for Recording Diet in Free-living UK Adults (SODIAT-2 Study)
Acronym: SODIAT-2
Status: Recruiting | Type: Observational
Sponsor: University of Reading (Other)
Collaborators: Aberystwyth University (Other); University of Cambridge (Other); Imperial College London (Other)
Responsible Party: Principal Investigator, Julie Lovegrove, Professor, University of Reading
Other Study IDs: UREC 24/43; (MR/W028336/1) (Other Grant/Funding Number: Medical Research Council (MRC) and the Biotechnology and Biological Sciences Research Council (BBSRC))
Record Dates: First submitted 2025-02-24; First posted 2025-03-17 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-07

CONDITIONS: Dietary Intake Assessment; Food Intake Measurement
Keywords: Nutrition; Health; Dietary reporting; Misreporting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine and blood samples will be retained. Dried capillary blood samples will be retained at the UoC but will not be used to extract DNA. They will be analysed for biomarkers of food/drink intake (e.g. fats and dairy products). Urine samples will be processed and retained in an acellular form (ensuring they are not relevant for DNA extraction) at the AberU. A range of biomarkers of food /drink intake will be measured at the end of study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Free-living adults living in GB: The study aims to recruit 133 adults living in GB with BMI more than 18.5 kg/m2 who are fluent in English. Participants will monitor their usual dietary intake during two 3-day monitoring periods during weeks 1 and 5 by wearing camera technology, self-collecting blood and urine samples at designated times, and completing online food frequency questionnaire on multiple occasions. During the calibration week (week 3) participants will consume the same 3-day test diet (either the diet for meat/fish consumers or non-consumers, as identified at screening).
  Interventions: Other: Measuring dietary intake

INTERVENTIONS:
Other: Measuring dietary intake — During 5-week study, participants will monitor their usual dietary intake during two 3-day periods (on weeks 1 and 5). During week 3 (calibration week) participants will consume a test diet. Wearable camera technology, self-collected blood and urine samples, and online FFQ (eNutri) will be used to monitor food intake during study weeks. Study tools as well as foods/drinks for the test diet will be delivered to each participant and they will be asked to comply with the study procedures in their home or working environment. Participants will post study samples and the study equipment/logs at designated times using pre-paid envelopes or a courier collection, respectively.

SUMMARY:
The aim of the SODIAT-2 study is to evaluate the effectiveness of dietary intake assessment tools in a real-world setting. These tools include wearable cameras, spot urine samples, capillary blood samples, and a web-based food frequency questionnaire (FFQ). The main questions it aims to answer are:

Is the accuracy of dietary assessment improved in free-living environments when a combination of subjective and objective assessments tools are used?

Secondary research questions are:

Can wearable cameras accurately monitor the daily dietary intake of free-living individuals? Does a combination of capillary blood samples and spot urine samples provide a robust assessment of the nutrient status and habitual dietary exposure in a free-living setting? Can data-driven integration of multiple emerging technologies create a dietary assessment tool that is low burden, accurate and scalable in free-living populations? Can a condensed FFQ estimate diet quality as effectively as a detailed FFQ?

Participants will:

Use the dietary assessment tools (wearable camera, spot urine, capillary blood, and eNutri FFQ web-app) as instructed over a 5-week period from their home and/or working space.

Take part in two monitoring weeks (week 1 and week 5) where they will record their usual dietary intake over 3 days.

Consume an identical 3-day study meal plan during the test (calibration) diet week 3, whilst repeating the monitoring week measurements.

This study aims to recruit 133 adults living in Great Britain (GB) to better understand how these tools perform outside of a clinical environment.

DETAILED DESCRIPTION:
The SODIAT project is a collaborative effort involving Aberystwyth University (AberU, project lead), University of Reading (UoR), Imperial College London (Imperial), and the University of Cambridge (UoC). Study 1, completed in July 2024, assessed the effectiveness of objective and subjective dietary intake assessment methods in highly-controlled clinical trial (protocol published at https://doi.org/10.12688/f1000research.155683.1) and informed the design of study 2.

Study 2 is led and sponsored by UoR. All study activities will be conducted remotely, with participants taking part from their usual locations (e.g., home, work).

►Screening and Welcome Week

Participants will use the online REDCap research platform to provide informed consent and complete a screening questionnaire to determine eligibility. Eligible participants will be contacted by a study researcher to discuss the study requirements, confirm consent, and schedule the study period.

A week before starting the 5-week study (Welcome Week), participants will be sent study materials/equipment and will be referred to the SODIAT webpage to view online video tutorials and read user guidelines for each study tool. Afterwards, participants will attend a video call with a study researcher to familiarize them with the study protocol and provide an opportunity to ask questions.

During the Welcome Week, participants will also self-collect a baseline blood sample (pre-video call) and complete the online eNutri FFQ to assess habitual diet. Within 2 days, they will then complete a condensed version of the FFQ to evaluate its effectiveness in estimating diet quality with reduced participant burden.

►5-week study period

Participants will follow their usual diet during weeks 1 & 5 and record their diet using study tools (wearable cameras, blood samples, urine samples and online FFQ) for 3 consecutive days (Monitoring Weeks). During week 3 (Calibration Week), participants will use the same study tools as before whilst consuming the 3-day test diet. There will be two test diets (one diet for meat/fish consumers and another slightly adapted for non-consumers), consisting of foods and drinks that are common in the UK. During this controlled part of the study, participants will be requested to eat/drink all foods and drinks provided (delivered by an online supermarket) but cannot consume anything extra. They will receive recommendations on serving sizes for each food/drink but participants can choose how much they eat (either more or less).

►Wearable cameras

Participants will wear a small camera unit mounted on glasses (or attached to their own frames) during the 3-day periods of weeks 1, 3, and 5 (days 1-3; 15-17 and 32-34). The camera automatically captures still images every 7 seconds to document food and drink intake. The camera will be worn from waking to going to bed, although participants will be instructed to remove the camera during private times (e.g., bathroom), sensitive locations (e.g., changing rooms, GP surgeries) and if unsafe to wear (e.g., driving), and log these occasions, as well as the camera start time, on a paper-based log. At the end of the study, encrypted SD cards containing the images will be returned to the research team at Imperial for secure processing.

Images will be pre-processed using AI to exclude irrelevant images, and blur identifying details (e.g., faces, device screens). Only anonymised images will be analysed by researchers to estimate dietary intake.

►Capillary blood samples

When fasted, participants will self-collect blood samples using OneDraw kits on day 4 of each study week (day 4, 18 and 35), which collect a few drops of blood from the upper arm/thigh onto a filter paper cartridge. A baseline sample will also be collected during the Welcome Week. Instructions and video tutorials will be provided, and samples will be mailed to researchers at UoC for storage and biomarker analysis.

►Spot urine samples

Over 4 consecutive days of each study week (days 1-4, 15-18, 32-35), participants will collect first morning void and last evening void urine samples using straw and vacuum tube kits. Samples will be temporarily stored in a refrigerator before mailing them to AberU for processing where biomarkers of food and drink intake will be analysed.

►Online FFQ (eNutri)

Participants will complete the online eNutri FFQ on six occasions. Both the original (long-format) and condensed FFQ will be completed during Welcome Week to capture habitual intake during the previous 4 weeks. During the study, a 3-day, condensed FFQ adapted to capture foods/drinks not well-represented by biomarker analysis, will be completed at the end of each recording week (day 4, 18 and 35). During the test diet week, the original FFQ, adapted to capture 3-day intakes, will also be completed (day 18). The FFQ inputs, nutrient and food group intakes, and diet quality data will be exported in pseudonymised format for analysis.

At the study's conclusion, participants will complete a short, online usability questionnaire about the study tools via REDCap (day 35).

Participants will mail their blood and urine samples at designated timepoints using pre-paid postage, and return all study equipment and logs at the end of the study via a courier collection.

Researchers will monitor adherence and communicate with participants as needed. Daily reminders will also be sent via email or text (SMS) message during the recording days.

► Statistical analysis

Accuracy of integrating multiple dietary assessment technologies to report dietary intake in free living environments will be measured during the calibration week (week 3) using dietary intake data collected from wearable cameras, spot urine samples, capillary blood samples, and self-reported FFQs.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Lives in Great Britain (England, Schotland and Walse)
* Able to read/understand instructions written in English and are fluent in English

Exclusion Criteria:

* Diagnosed or self-report as being underweight (have a body mass index (BMI) of less than 18.5 kg/m2)
* Are unwilling/unable to collect urine and blood samples, use the wearable camera as instructed and/or spend 20-30 min online recording what they've recently had to eat/drink on multiple occasions
* Are unwilling/unable to have a video call with a researcher with cameras turned on
* Are unwilling/unable to post samples on specific days and receive/send a larger parcel at the start/end of the study (note: all return packaging and postage will be provided by us and will include a courier delivery and collection)
* Are unwilling/unable to receive a single grocery delivery from Sainsbury's or Tesco online supermarkets (delivery to be arranged by us), includes living in a postcode area that cannot receive grocery deliveries from Tesco or Sainsburys as well as not having space to refrigerate and freeze items.
* Are unwilling/unable to eat/drink any items on the calibration menu, e.g., food allergies/intolerances, dislike of food items, unable eat (e.g. vegan or have to avoid for a medical condition) or cannot eat 3 meals plus snacks daily (note: vegetarians can take part)
* Are unwilling/unable to avoid taking dietary and herbal supplements for at least 1 week before and during the 5-week study (e.g. fish oils, vitamins, iron, protein shakes, nutrient powders, joint care)
* Are pregnant, may be pregnant or breast-feeding
* Currently experiencing, recovering or at a high risk of an eating disorder (e.g., previous diagnosis, or concerns that you have an unhealthy relationship with food)
* Have a health condition, are taking medication and/or undergoing medical treatment that affects metabolism, appetite and/or ability to eat the calibration menu (e.g. cancer, chemotherapy, diabetes, gastrointestinal disorders (such as inflammatory bowel disease, Crohn's disease), kidney disease, liver disease, HIV or AIDS)
* Are taking any of the following medications: androgens, blood thinners, phenytoin, erythromycin, or thyroid hormones
* Long-term use of any of the following medications: anti-inflammatories (NSAIDS), steroids/corticosteroids or antibiotics (eligible following a 4-week washout after short term use; eligible if use is infrequent)
* Use illicit substances/recreational drugs
* Have been diagnosed with dementia or other conditions affecting memory
* Do not have anyone at home, work, etc. to help them if they require assistance to use the study tools (such as arthritis, Parkinson's disease, sight loss, etc.)

If the participants have recently taken part in another intervention study, a 4-week washout will be required before they are able to start the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: UK population.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Dietary intake measured by wearable camera technology. | Days 1- 3 (week 1), days 15-17 (week 3) and days 32-34 (week 5).
  Wearable cameras will be worn by the participants during the study days. Images from wearable cameras will be analysed to estimate what foods and drinks were consumed during the study days, as well as estimating their portion sizes (grams per day).
Dietary intake measured by spot urine. | Morning and evening spot urine samples collected over 4 consecutive days on weeks 1, 3 and 5 (days 1-4, 15-18, 32-35).
  A range of biomarkers indicating what a person has eaten/drank will be measured in urine samples.
Dietary intake measured by blood sample. | Samples collected at fasted state in the morning of days 4, 18 and 35 (weeks 1, 3 and 5).
  A range of food/drink biomarkers will be measured in capillary blood samples to indicate what a person has eaten/ drank.
Monitoring/calibration week dietary intake (condensed 3-day FFQ). | Days 4, 18 and 35 (weeks 1, 3 & 5).
  Food/drink intake during the 3-day study periods will be measured by the 3-day condensed FFQ (adapted to capture foods not represented by biomarker analysis). Outcomes include dietary intakes (frequency, portion size and grams per day) for each FFQ item, nutrient intakes, food group intakes and diet quality score.

SECONDARY OUTCOMES:
Habitual dietary intake (original eNutri FFQ). | Baseline.
  Habitual intake will be measured by the original 4-week eNutri FFQ. Outcomes include dietary intakes (frequency, portion size and grams per day) for each FFQ item, nutrient intakes, food group intakes and diet quality score.
Habitual dietary intake (condensed original FFQ). | Baseline, after original eNutri FFQ.
  Habitual intake will be measured by the condensed 4-week eNutri. Outcomes include dietary intakes (frequency, portion size and grams per day) for each FFQ item, nutrient intakes, food group intakes and diet quality score.
Calibration week dietary intake (3-day eNutri FFQ). | Day 18, week 3.
  Food/drink intake during the 3-day calibration week ( week 3) will be measured by the 3-day FFQ. Outcomes include dietary intakes (frequency, portion size and grams per day) for each FFQ item, nutrient intakes, food group intakes and diet quality score.
Usability questionnaire for each research tool. | Day 35, week 5.
  Short qualitative feedback questionnaire will be administered online via REDCap to determine participants' perspectives on usability of each study tool (including Likert scale questions "strongly disagree to strongly agree" and free text responses).

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Beckmann, Dr, Principal Investigator — Department of Life Sciences, Aberystwyth University; Julie A Lovegrove, Professor, Principal Investigator — Hugh Sinclair Unit of Human Nutrition Department of Food and Nutritional Sciences, University of Reading; Gary Frost, Professor, Principal Investigator — Nutrition Research Section, Hammersmith Hospital Campus, Imperial College
Locations (4):
- United Kingdom (4):
  - Hugh Sinclair Unit of Human Nutrition, University of Reading, Reading, Berkshire
  - Department of Life Sciences, Aberystwyth University, Aberystwyth
  - University of Cambridge, Pathology building level 4, Addenbrooke's Hospital, Cambridge
  - Nutrition Research Section, Hammersmith Hospital Campus, Imperial College, London

IPD SHARING:
Plan to Share IPD: Yes
Anonymised individual participant data will be shared in accordance with confidentiality and consent agreements. This may include: sociodemographic information, anthropometric measurements, dietary intake data, blood and urine biomarkers. Public data repositories (to be agreed by the project team) will be used preserving fully anonymised individual data.
Supporting Information: Study Protocol, ICF
Time Frame: To be made available at the point of publication.
Access Criteria: The SODIAT Project Lead, Dr Manfred Beckmann (AberU) will have overall authority over the central data repository. The Principal Investigator at UoR, Professor Julie Lovegrove, will have authority over any data collected and stored at UoR, including REDCap and eNutri.

REFERENCES:
- See also: SODIAT webpage — https://sodiat.org/